CLINICAL TRIAL: NCT04017351
Title: Virtual Assistant for Plastic Surgery Patients - Impact on the Clerical Burden, Resource Utilization, Patient and Provider Satisfaction, and Patient Surgical Outcomes.
Brief Title: Virtual Assistant for Plastic Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Antonio J. Forte, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-001980
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Surgery
Keywords: Plastic; Virtual Assistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with virtual assistance (Experimental): Subjects receiving current standard of care for a surgical procedure within the department of plastic surgery will have access to artificial intelligence virtual assistance (AIVA)
  Interventions: Other: Artificial Intelligence Virtual Assistant
- Subjects without virtual assistance (No Intervention): Subjects receiving current standard of care for a surgical procedure within the department of plastic surgery

INTERVENTIONS:
Other: Artificial Intelligence Virtual Assistant — Virtual assistance application for subjects to ask questions and get information regarding planned surgery
  Other Names: AIVA
  Arms: Subjects with virtual assistance

SUMMARY:
Researchers are trying determine the long term impact when patients have access to the artificial intelligence virtual assistant (AIVA) as a complimentary resource.

DETAILED DESCRIPTION:
Eligible subjects will be randomized into to two groups. One group of subjects will be given access to the AIVA will be instructed to ask, at home, questions regarding the planned surgery to the AIVA application on their mobile phone. The other group will be instructed to call to the Standard of Care call center with questions related to their treatments. Researchers will follow up with all subjects from both groups for a 1 year amount of time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects above 18 years old
* Able to use applications on mobile phones and consent to participate
* Adult subjects in the Plastic Surgery outpatient clinic of Mayo Clinic Florida

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of phone calls | 12 months
  The total number of phone calls from subjects
Duration of phone call | 12 months
  Length of phone calls from subjects. Measured in minutes
Nature of phone call | 12 months
  The total number of phone calls related to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials